CLINICAL TRIAL: NCT03712462
Title: Improving Weight Loss Outcomes for Binge Eating Disorder.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Yale University (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1803006178; R01DK117072 (NIH)
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Eating Disorder; Binge-Eating Disorder; Weight Loss; Binge Eating
Keywords: Eating Disorder; Binge Eating; Binge Eating Disorder; Weight Loss
MeSH Terms: conditions — Feeding and Eating Disorders; Binge-Eating Disorder; Weight Loss; Bulimia | interventions — Beds

STUDY DESIGN:
Intervention Model Description: The novel acceptance-based behavioral weight loss therapy is being compared to standard behavioral weight loss therapy for individuals with binge eating disorder.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABBT Weight Loss Therapy for BED (Experimental): Acceptance-Based Behavioral Weight Loss Therapy for BED
  Interventions: Behavioral: Acceptance-Based Behavioral Weight Loss Therapy for BED
- Standard Behavior Therapy (Active Comparator): Standard Behavioral Weight Loss Therapy
  Interventions: Behavioral: Standard Behavior Therapy

INTERVENTIONS:
Behavioral: Acceptance-Based Behavioral Weight Loss Therapy for BED — ABBT group therapy incorporates standard behavioral and acceptance-based strategies and was adapted to meet suit the unique needs of BED.
  Arms: ABBT Weight Loss Therapy for BED
Behavioral: Standard Behavior Therapy — SBT group therapy will be adapted from the gold-standard standard behavioral therapy manuals used from previous weight loss studies.
  Arms: Standard Behavior Therapy

SUMMARY:
This study aims to develop and evaluate the efficacy of a behavioral weight loss treatment approach for individuals with binge eating disorder to both reduce their binge eating behaviors and lose weight.

DETAILED DESCRIPTION:
In the current study, we propose to (a) compare the efficacy of an acceptance-based behavioral treatment (ABBT) that targets both binge eating and weight loss in patients with binge eating disorder (BED) to a Standard Behavioral Weight Loss Treatment (SBT), (b) evaluate the extent to which ABBT and SBT target shared maintenance factors for binge eating and overeating episodes, and (c) assess whether treatment efficacy is moderated by baseline values of constructs targeted in ABBT. Our study will be the first to evaluate an ABBT for BED designed to 1) address maintenance factors that give rise to both binge eating episodes and overeating episodes without loss of control and 2) increase adherence to BWL prescriptions.

ELIGIBILITY:
Inclusion Criteria:

* Meet the DSM-5 criteria for Binge Eating Disorder
* Have a BMI range of 27-50kg/m2

Exclusion Criteria:

* are unable to fluently speak, write, and read English
* are currently experiencing severe psychopathology that would limit their ability to engage in study (e.g., suicidality, substance use disorder, psychotic disorder)
* are unable to engage in moderate physical activity (i.e., walk 2 blocks without rest)
* have a medical condition (e.g., acute coronary syndrome, type I diabetes) that would pose a risk to the participant during intervention, cause a change in weight, or limit ability to comply with the recommendations of the program
* Pregnant or planning to become pregnant in the next 2 years
* Recently began a course of or changed the dosage of medication that can cause significant change in weight
* Have a history of bariatric surgery
* Have had weight loss of > 5% in the past 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Stratton Hall, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ABBT Weight Loss Therapy for BED | Standard Behavior Therapy
Started | 63 | 63
Completed | 43 | 43
Not Completed | 20 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABBT Weight Loss Therapy for BED | Standard Behavior Therapy | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.56 (12.41) | 51.05 (11.60) | 51.30 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Missing data for two participants from ABT and two participants from SBT.
  Participants
    number analyzed (Participants) | 61 | 61 | 122
    Female | 51 | 49 | 100
    Male | 10 | 12 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 58 | 54 | 112
  Unknown or Not Reported | 3 | 8 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 15 | 31
  White | 44 | 44 | 88
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 126
Baseline EDE Global Score [Mean (Standard Deviation); unit: scores on a scale] — Measure Description: The Eating Disorder Examination (EDE) is a diagnostic interview for the assessment of eating disorder symptoms, including binge eating frequency, compensatory behavior frequency, and global eating pathology. The EDE yields a global score and four subscale scores (Restraint, Eating concern, Shape concern, Weight concern), with higher scores indicating greater severity of eating disorder pathology. To obtain the global score, the subscale scores (which range from 0 to 6) are summed, and the resulting total is divided by the number of subscales (i.e. four).
  scores on a scale | 2.29 (0.68) | 1.72 (0.76) | 2.01 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Weight Loss
Description: Between-group changes in percent weight loss from baseline 1 month, 3 months, and 6 months into the study, at post-treatment (1 year after baseline) and at the one year follow-up assessment (2 years after the baseline).
Time Frame: Changes from baseline assessment (before beginning treatment), to post-treatment assessment (1 year after baseline assessment), to follow-up assessment (2 years after baseline assessment)
Measure: Mean (Standard Deviation); unit: percentage of weight loss
Arm/Group | ABBT Weight Loss Therapy for BED | Standard Behavior Therapy
Number analyzed (Participants) | 63 | 63
percentage of weight loss
  Baseline | 0 (0) | 0 (0)
  1 Month | -2.13 (3.68) | -2.15 (2.85)
  3 Months | -5.46 (5.41) | -5.25 (4.32)
  6 Months | -7.65 (7.37) | -6.97 (5.92)
  Post-Treatment | -7.46 (9.67) | -7.06 (7.42)
  1 Year Follow-Up | -4.76 (9.01) | -3.52 (7.02)

2. Secondary Outcome: Eating Disorder Examination Questionnaire
Description: The Eating Disorder Examination Questionnaire measures eating pathology. The EDE-Q yields four subscale scores: Restraint, Eating Concern, Shape Concern, and Weight Concern. The possible score range for each subscale is 0 to 6. The total score may also be reported (determined by averaging the subscale scores); the score range for the total score is also 0 to 6. For subscale scores and total score, higher scores indicate more severe pathology. The restraint sub-scale of the EDE-Q will be used to assess utilization of skills related to reducing dietary restraint.
  Assessing changes in EDE Global score.
Time Frame: Baseline, Post-Treatment (1 year after baseline), and 1 Year Follow-Up (2 years after baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ABBT Weight Loss Therapy for BED | Standard Behavior Therapy
Number analyzed (Participants) | 63 | 63
score on a scale
  Baseline | 2.29 (0.68) | 1.72 (0.76)
  Post-Treatment | 2.49 (0.77) | 1.49 (0.78)
  1 Year Follow-Up | 1.50 (0.70) | 1.60 (0.81)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | ABBT Weight Loss Therapy for BED | Standard Behavior Therapy
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 0/63 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-26): https://cdn.clinicaltrials.gov/large-docs/62/NCT03712462/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT03712462/SAP_001.pdf